CLINICAL TRIAL: NCT03121027
Title: Burden of Anemia Among Ever-married Women in Bangladesh
Brief Title: Burden of Anemia Among Ever-married Women in Bangladesh: Does Household Economic Inequality Matter?
Status: Completed | Type: Observational
Sponsor: Shahjalal University of Science and Technology (Other)
Responsible Party: Principal Investigator, G.M. Rabiul Islam, Associate Professor, Shahjalal University of Science and Technology
Other Study IDs: AW-FET
Record Dates: First submitted 2017-04-11; First posted 2017-04-19 (Actual); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Anemia
Keywords: Anemia; Ever married women; Economic inequality; Diabetes; Maternity; BMI
MeSH Terms: conditions — Anemia; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Despite significant advances in the field of medicine and healthcare, anemia continues to be a major public health problem worldwide. The situation is particularly acute in developing countries where females belonging to the reproductive age category are especially vulnerable to the malady. Given the multifactorial nature of this disease, correcting anemia often requires the adoption of an integrated approach. Therefore, it is imperative that the role played by the "causes of the causes" (i.e., the sociodemographic determinants of risk), along with other contributing factors, must be identified, and addressed in order to effectively combat this disease. In general, it is terrible to sort out the psychosocial factors from the demographics, environmental and poverty-related causes. Therefore, the objective of this study is to use a nationwide representative survey to explore the magnitude of household economic inequalities contribute towards the prevalence of anemia among ever-married women in Bangladesh. The study also aims to examine the inference of other explanatory variables that frequently had supposed decomposing on the burden of anemia. Thus, this study answers the questions: (a) what are the strengths and likelihoods of having mild, moderate or severe anemia among the ever married women of different SES?; (b) do other factors viz., demographics, diabetes, maternity, and BMI affects the strength and form of the association between SES and anemia?; (c) which explanatory variable is more prone to pose anemia among the women? As the burden of anemia is one of the key policy issues facing Bangladesh, the findings generated by this study are expected to contribute towards further policy making by virtue of identifying associated risk factors. This is expected to be instrumental for program purposes designed to prevent anemia among Bangladeshi women.

DETAILED DESCRIPTION:
This study was carried out with the approval of ICF International ( Address: 11785 Beltsville Drive Suite 300 Calverton, MD 20705 USA). The data from the 2011 Bangladesh Demographic and Health Survey (BDHS), conducted under the authority of the National Institute of Population Research and Training (NIPORT) of the Ministry of Health and Family Welfare of Bangladesh will be used for this study. Mitra and Associates, a Bangladeshi research firm located in Dhaka implemented the survey and ICF International of Calverton, Maryland, USA, arranged the technical support to the mission as the part of its international Demographic and Health Surveys database (MEASURE DHS). Procedures and questionnaires for standard DHS surveys have been reviewed and approved by the ICF International Institutional Review Board (IRB). (See more at: http://www.dhsprogram.com/What-We-Do/Protecting-the-Privacy-of-DHS-Survey-Respondents.cfm#sthash.qc30dbXO.dpuf) The data collection processes for the BDHS was executed as per the approval of the ORC Macro-institutional review board. The survey protocol was reviewed and approved by the National Ethics Review Committee of the Bangladesh Ministry of Health and Family Welfare. As per BDHS guidelines, informed consent was obtained from all respondents before starting the interview along with an oral clarification offered by the interviewers themselves. Respondents were well informed with regards to the intended use of the gathered data (assessment of health needs and planning health services), the voluntary nature of the study, potential risks of participation in the study, the confidentiality of answers/results of the individual interview and biomarker assay, and that the examination was free of cost. Prior to the blood collection and examination, participants were also well informed about the purpose of the study.

A stratified, multistage cluster sampling strategy was followed in order to construct a national representative household-based sample. To generate this, 600 primary sampling units (207 from urban areas and 393 from rural areas) were raised from the sampling frame created for the 2011 Bangladeshi census. From each primary sampling unit, households were nominated randomly and 17,964 households were selected for interview. Face-to-face interviews were effectively completed among 17,141 selected households. Finally, in these households a total of 18,222 ever married women age 12-49 were identified and 17,842 were interviewed successfully. A total of 5920 ever-married women aged between 15-49 years who resided in one-third of the randomly selected households were selected as subjects for the biomarker assay for anemia study.

ELIGIBILITY:
Inclusion criteria:

* Ever-married women: Those who get married, divorced and the widow is also included.
* Exclusion criteria:

Not married women: Those who never married.

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Ever married Women in Bangladesh
Sampling Method: Non-Probability Sample
Enrollment: 5920 (Actual)
Dates: Start 2011-05-11 (Actual); Primary Completion 2011-07-08 (Actual); Study Completion 2012-01-18 (Actual)

PRIMARY OUTCOMES:
Anemia | Baseline
  Hemoglobin concentration will be used as the parameter for diagnosing anemia. For the purpose of this study, "anemia" will be defined as per WHO, 2011 guidelines for the diagnosis of anemia. Briefly, in the case of pregnant women, a hemoglobin concentration of less than 70 g/L will be used to define severe anemia, between 70-99.99 g/L will be used for defining moderate anemia while 100-109.99 g/L will be consider to correspond to mild anemia (n=372). In non-pregnant women, a hemoglobin concentration of less than 80 g/L will be used to define severe anemia, 80-109.99 g/L for moderate anemia, and 110-119.99 g/L to correspond to mild anemia. In accordance with the recommendation of the Center for Disease Prevention of United States, and in agreement with the World Health Organization, the blood assay report for anemia will be adjusted for altitude and smoking during the categorization into "severe" "moderate" or "mild" anemia.

CONTACTS AND LOCATIONS:
Overall Officials: GM R. Islam, PhD, Principal Investigator — Shahjalal University of Science and Technology
Locations (1):
- Data analysis, Sylhet, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- Available data/document: Individual Participant Data Set — https://dhsprogram.com/pubs/pdf/fr265/fr265.pdf — Detail about sampling and BDHS 2011 report